CLINICAL TRIAL: NCT01749501
Title: Premedication for Non-Emergency Endotracheal Intubation In the NICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Martin Espinosa, MD (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor-Investigator, Martin Espinosa, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-271
Record Dates: First submitted 2012-09-28; First posted 2012-12-13 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rocuronium (Active Comparator): 0.6 mg/kg once
  Interventions: Drug: Rocuronium
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rocuronium — 0.6 mg/Kg once
  Other Names: Zemuron
  Arms: Rocuronium
Other: Placebo — Normal saline same amt as 0.6mg/kg of study drug
  Arms: Placebo

SUMMARY:
Those infants who received the muscle relaxation in combination with the vagolytic (reduce vagus nerve impulses) and pain medication will have reduced time to successful intubation (placement of tube into the lungs), a decrease in the number of attempts, and better intubation conditions reported by the practitioner. The objectives of the study include: 1.) Does the medication protocol outlined in this study provide optimal intubation conditions? (i.e.good jaw relaxation, open and immobile vocal cords and suppression of gag reflex) 2.) Does the addition of a muscle relaxant prior to intubation contribute to less attempts and achieving successful intubation as opposed to neonates who do not receive the muscle relaxant.

DETAILED DESCRIPTION:
The investigators project will study two different strategies of pre-medication in an attempt to eliminate the pain and discomfort associated with the elective intubation procedure. The study will be blinded and patients will be randomized in two different arms according to gestational age and identified by study number for pre-medication protocols. Demographic as well as study information prior, during and post intubation attempt will be recorded and closely monitored. Each patient will be monitored for study purposes for at least 24 hours after intubation attempt to record any potential side effects of the medication. The investigators plan to have a data safety monitoring board established composed of three pediatric doctors / specialists not associated with this study.

The response of paralysis, onset and duration will be assessed clinically. Onset of muscle relaxation will be described as the absence of spontaneous movements and flaccidity, measured in seconds from the end of the medication administration. Duration of paralysis will be determined by the difference in time from the onset of paralysis to the return of spontaneous movements and pre-intubation tone

ELIGIBILITY:
Inclusion criteria:

1. Infants admitted to the NICU at Beaumont Children's Hospital Royal Oak and Troy.
2. Gestational Age 28 0/7 weeks (or post menstrual age 28 0/7 weeks) or higher
3. Infants who require endotracheal intubation on a non-emergent basis
4. Signed informed consent by parents

Exclusion criteria:

1. intubations that occurred in the delivery room or for other emergent basis,
2. absence of intravenous access
3. abnormality of the airway
4. known or family history of neuromuscular disorder
5. renal insufficiency (urine output <0.6 mL/kg per hour or creatine >1.7 mg/dL if > 1 day of age)
6. known hepatic insufficiency (abnormal liver function or coagulation laboratory results)
7. Current diagnosis of pulmonary hypertension
8. Any infant deemed by the attending neonatologist as unstable or unfit for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Espinosa, MD, Principal Investigator — Corewell Health East

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 69 participants consented but only 45 needed the study procedure
Period: Overall Study
Arm/Group | Rocuronium | Placebo
Started | 22 | 23
Completed | 22 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocuronium | Placebo | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 23 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: post menstrual age (PMA) weeks] | 35.4 (4.47) | 33.88 (3.65) | 34.62 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Present the Percentage of Participants With an Excellent Ease of Intubation Rating
Description: percentage of participants with an excellent ease of intubation rating based on Scale of 1-4 (1 Being Excellent, 4 Being Poor),"
Time Frame: 24 hours after intubation period
Measure: Number; unit: % reported as excellent
Arm/Group | Rocuronium | Placebo
Number analyzed (Participants) | 22 | 23
% reported as excellent | 91 | 17

2. Secondary Outcome: Timing of Entire Procedure (Stopwatch)and Recording Number of Attempts to Successful Intubation Recorded.
Time Frame: 24 hours after intubation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rocuronium | Placebo
Number analyzed (Participants) | 22 | 23
minutes | 2.94 (5.0) | 4.95 (5.43)

ADVERSE EVENTS:
Arm/Group | Rocuronium | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No